CLINICAL TRIAL: NCT06770686
Title: Development of Nursing Care Bundle for the Prevention of Pressure Injuries, the Impact on the Rate and Cost of Pressure Injuries
Brief Title: Development of a Nursing Care Bundle to Prevent Pressure Injuries and Its Impact on Rates and Costs
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2024.066.IRB2.039
Record Dates: First submitted 2025-01-07; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Pressure Injury; Hospital Acquired Pressure Ulcer
Keywords: Care Bundles; Cost
MeSH Terms: conditions — Pressure Ulcer | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Care (Active Comparator): Patients in the control group will receive routine care related to pressure injury prevention administered by the institution. Routine care includes standard interventions such as checking pressure points at twice-daily shift changes, positioning every 2 hours, skin assessment, and wound assessment.
  Interventions: Other: Control Group
- Care Bundle Group (Experimental): A nursing care bundle will be applied to patients in the intervention group. The implementation status of the nursing interventions included in the care bundle for each patient will be observed by the researcher and recorded on the "Care Bundle Observer Form." Recording of the applications performed on the monitoring form will be encouraged.
  Interventions: Other: Intervention Group

INTERVENTIONS:
Other: Intervention Group — A nursing care bundle will be applied to patients in the intervention group. The implementation status of the nursing interventions included in the care bundle for each patient will be observed by the researcher and recorded on the "Care Bundle Observer Form." Recording of the applications performed on the monitoring form will be encouraged.
  Other Names: Maintenance bundle care group
  Arms: Care Bundle Group
Other: Control Group — They will receive standard care
  Arms: Standard Care

SUMMARY:
Pressure injuries (PIs) represent a significant clinical complication for patients worldwide and pose financial and quality challenges for healthcare systems. These wounds, which are highly challenging to treat and care for both patients and caregivers, lead to physical and psychological trauma, negatively affect daily life activities, reduce quality of life, and increase care costs (Padula et al., 2019; Yilmazer & Tüzer, 2022). Moreover, the expenses associated with treatment are 2.5 times higher than those for prevention (Lyder & Ayello, 2007). Additionally, they often prolong hospital stays and increase the time nurses spend on care (Yilmazer & Tüzer, 2022).

According to the National Pressure Injury Advisory Panel (NPIAP, 2019), providing high-quality care for patients with PIs requires adopting a multidisciplinary, standardized care approach tailored to the specific needs of patients (Heasler, 2019). Past and current literature supports the use of evidence-based care bundles to reduce PIs (Coyer et al., 2015; Chaboyer et al., 2015; Amr et al., 2017; Deakin et al., 2020; Yilmazer & Tüzer, 2022; Wang et al., 2023). A care bundle is a critical element for standardizing and enhancing the quality of nursing care through the utilization of evidence-based clinical practice guidelines by healthcare professionals. Therefore, adopting these evidence-based approaches will improve the consistency and quality of nursing care, enhance patient outcomes, and reduce institutional costs. Moreover, the use of care bundles during interventions promotes teamwork and collaboration while supporting the development of a common language (Anderson et al., 2015; Institute for Healthcare Improvement, 2021).

This study aims to reduce PIs, enhance the quality of patient care, lower healthcare costs, and improve overall patient outcomes through the development and implementation of a nursing care bundle based on evidence in the literature. The widespread use of the care bundle, grounded in achieved outcomes, will contribute to the prevention of PIs. Additionally, it will serve as a supportive tool for nurses to improve the quality of care.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older
* Patients who fall into all risk categories assessed by the Braden scale
* Not having developed a pressure injury anywhere on their body
* Expectation of a minimum of 24 hours or more in the intensive care unit

Exclusion Criteria:

* Being 18 years of age or younger
* Having and developing a pressure injury anywhere on their body
* Expectation of a less than 24-hour stay in the intensive care unit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Hospital-acquired pressure injuries rate | For 3 months

SECONDARY OUTCOMES:
Cost analysis results | For 3 months

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang LP, Gao MM, Wang XQ, Gu MM, Qi QD. Effects of bundle-care interventions on pressure ulcers in patients with stroke: A meta-analysis. Int Wound J. 2023 Oct 18;21(2):e14432. doi: 10.1111/iwj.14432. Online ahead of print. PMID 37853846
- [Background] Coyer F, Gardner A, Doubrovsky A, Cole R, Ryan FM, Allen C, McNamara G. Reducing pressure injuries in critically ill patients by using a patient skin integrity care bundle (InSPiRE). Am J Crit Care. 2015 May;24(3):199-209. doi: 10.4037/ajcc2015930. PMID 25934716